CLINICAL TRIAL: NCT07180238
Title: Concept Elicitation and Patient Experience Mapping in Sepsis-associated Acute Kidney Injury
Brief Title: Concept Elicitation and Patient Experience Mapping in SA-AKI
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTIN816B12002
Record Dates: First submitted 2025-09-10; First posted 2025-09-18 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Sepsis-associated Acute Kidney Injury
Keywords: Sepsis; Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a concept elicitation study on patient's experiences of Sepsis-associated Acute Kidney Injury (SA-AKI)

DETAILED DESCRIPTION:
The purpose of this study is to elicit concepts of interests in patients who experienced SA-AKI. The study also aims to map experiences from patient and caregiver perspectives, including treatment pathways and barriers to SA-AKI treatment, the burden of SA-AKI and unmet needs, and the disease's humanistic, societal, and economic impacts. This study is a cross-sectional, non-interventional qualitative interview study of up to 30 people who have experienced SA-AKI from the US and Germany. Participants will be screened for eligibility, provide consent, and complete a virtual, hybrid 60-minute semi-structured concept elicitation (CE) and patient experience interview. Transcripts will be reviewed by analysts and analysed according to a qualitative analysis plan including a thematic analysis of the coded transcripts. This is a minimal risk study. All information will be kept confidential, and information will be stored on a secure network which is only accessible to the study team.

ELIGIBILITY:
Inclusion Criteria:

Potential participants who were diagnosed with SA-AKI (KDIGO stage I, II or III) must meet the following eligibility criteria:

* ≥18 to ≤ 85 years of age
* First diagnosis of SA-AKI at least 6 months prior to screening date, but no more than 10 years
* Admitted due to sepsis and/or AKI to intensive care unit (ICU), intermediate care unit (IMCU), or high-dependency care unit, or developed sepsis and/or AKI during their inpatient hospital stay.
* Resident of country of study (US or Germany)
* Access to computer, tablet, or smartphone with internet connection
* Willing to participate in an audio recorded interview

Participants will be required to present confirmation of diagnosis (COD) rather than relying on a self-reported diagnosis. Sepsis and AKI diagnoses will be confirmed through one of the following:

* Copy of medical records (e.g., portable document format [PDF] file of electronic health record)
* Physician confirmation of diagnosis of sepsis and AKI (post-sepsis)

Potential caregiver participants must meet the following criteria:

* ≥18 to ≤ 85 years of age
* Primary caregiver/care-partner for eligible participant who experienced SA-AKI
* Resident of country of study (US or Germany)
* Access to computer, tablet, or smartphone with internet connection
* Willing to participate in an audio recorded interview

Exclusion Criteria:

Potential participants are not eligible if they meet any of the following criteria:

* Less than age of majority in locality (Participant is not considered an adult in their country or region)
* Not willing to participate in an audio recorded interview
* Not able to participate in the interview or complete required study surveys, based on the discretion of the study team

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have experienced SA-AKI. A subset of the interviews (50%-70%) will include a caregiver/care-partner in a dyad interview (a type of interview that involves two respondents). In addition, the study team targets for a minimum of 50% of participants that have been diagnosed with SA-AKI no longer than 5 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Patient perspective on sign, symptoms and impacts of SA-AKI | Up to 3 months
  A 60-min qualitative interview will be conducted and transcripts will be coded to assess which signs, symptoms and impacts of SA-AKI have been experienced by the participant

SECONDARY OUTCOMES:
Patient experiences on treatment pathways and barriers to SA-AKI treatment, the burden of SA-AKI and unmet needs, and the humanistic, societal, and economic impacts | Up to 3 months
  A 60-min qualitative interview will be conducted and transripts will be coded to assess the treatment pathways and barriers to SA-AKI treatment, the burden of SA-AKI and unmet needs, and the humanistic, societal, and economic impacts

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No